CLINICAL TRIAL: NCT05050396
Title: Comparison of The Effect of Cooled Versus Thermocoagulant Radiofrequency Ablation on Pain Relief of Knee Osteoarthritis
Brief Title: Radiofrequency Ablation on Pain Relief of Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Saif Eldeen Gamal Khalaf, Assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pain relief of osteoarthritis
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooled radio frequency (Experimental): In CRF, water circulates inside the probe to remove heat, modulating the thermal heat in the tissue to around 60°C, and alters the overall size, shape, and projections of lesions compared to conventional RFA. It is postulated that the greater sized CRF lesions may reduce the number of technical failures in the setting of a complex and variable neuronal innervation to the knee. The ability to target a greater amount of neuronal tissue is believed to produce long-term pain relief at least to the duration of relief produced by conventional RFA [27]
  Interventions: Procedure: Cooled versus thermocoagulant Radiofrequency Ablation in pain relief of knee osteoarthritis
- Thermocoagulant radio frequency (Experimental): Conventional radiofrequency Ablation RFA of the knee can be performed under fluoroscopic, or other imaging, guidance, with a cannula advanced into the joint towards the area connecting the shaft to the epicondyle. The area is stimulated to identify the nerve position and to ensure that no motor nerves are activated, as evidenced by absence of fasciculations. The RF electrode is then advanced through the cannula to the target area [18] The electrode tip heats up targeted local tissue within a few millimeters to a temperature typically greater than 47°C (ranging from 70°C to 90°C) for 120 130 seconds, generated through an electromagnetic field with a frequency of 250 kHz . [15,18] The ablative heat is provided via flow of electrical current, generating a well-delineated lesion [24]
  Interventions: Procedure: Cooled versus thermocoagulant Radiofrequency Ablation in pain relief of knee osteoarthritis

INTERVENTIONS:
Procedure: Cooled versus thermocoagulant Radiofrequency Ablation in pain relief of knee osteoarthritis — Radiofrequency (RF) ablation, or modulation of the sensory innervation surrounding the knee, specifically the genicular nerves (GNs), has emerged as a therapeutic option to treat chronic knee OA pain for patients who are unresponsive to conservative treatments or are unsuitable candidates for total knee arthroplasty (TKA). [16, 17] Similar to conventional RFA, water-cooled radiofrequency (CRF) ablation is a novel technology that utilizes thermal ablative mechanisms; however, CRF gives the ability to create a greater local neuronal lesion to increase the changes of effective denervation [20]

SUMMARY:
Introduction

Osteoarthritis (OA) is a chronic, progressive disease with high disability and teratogenicity in the joints. Deterioration of the articular cartilage is the main problem associated with osteoarthritis, which decreases joint space between the two bones[1].

Clinically, patients with knee OA typically present with a chief complaint of pain, often associated with limited range of motion, stiffness, osteophytes, crepitus, and effusions. Due to the progressive degenerative nature of OA and the associated pain, patients become more physically impaired through the course of the disease [6].

One of the main tissues affected by this disease is the articular cartilage, which is a thin tissue covering the bony end in the joint that mainly provides mechanical support and lubrication during joint movement [7].

Age, previous knee injuries, but also obesity(increased body mass index(BMI)) ,joint malalignment and instability that result in increased mechanical stress are all strong risk factors for the development of knee OA [8-10].

Magnetic resonance imaging (MRI), arthroscopy examination, high-frequency color ultrasound and thermal texture maps are the four most acceptable types of imaging examinations. These examinations cannot only help diagnose KOA, but they can also assess the severity of joint damage and evaluate disease progression and treatment [11,12].

Treatment options for patients with OA include: conservative approaches, such as weight loss, physical therapy, and pharmacological interventions, while the more invasive approaches include intraarticular injections, joint preserving surgical treatment, and total knee arthroplasty (TKA). [13, 14] Radiofrequency ablation (RFA) is a novel technique that also recently gained popularity in alleviating chronic pain in patients with musculoskeletal disorders such as OA [15] Radiofrequency (RF) ablation, or modulation of the sensory innervation surrounding the knee, specifically the genicular nerves (GNs), has emerged as a therapeutic option to treat chronic knee OA pain for patients who are unresponsive to conservative treatments or are unsuitable candidates for total knee arthroplasty (TKA). [16, 17]

DETAILED DESCRIPTION:
Introduction

Osteoarthritis (OA) is a chronic, progressive disease with high disability and teratogenicity in the joints. Deterioration of the articular cartilage is the main problem associated with osteoarthritis, which decreases joint space between the two bones[1].

Because of the higher prevalence of asymptomatic OA, it is approximated that 250 million people all over the world suﬀer from OA [2,3].

The prevalence of knee OA increased signiﬁcantly over the last decades and continues to rise, partially because of the increasing prevalence of obesity and other risk factors, [4].

It is estimated that the prevalence of knee OA among adults 60 years of age or older is approximately 10% in men and 13% in women [5].

Clinically, patients with knee OA typically present with a chief complaint of pain, often associated with limited range of motion, stiffness, osteophytes, crepitus, and effusions. Due to the progressive degenerative nature of OA and the associated pain, patients become more physically impaired through the course of the disease [6].

One of the main tissues affected by this disease is the articular cartilage, which is a thin tissue covering the bony end in the joint that mainly provides mechanical support and lubrication during joint movement [7].

Age, previous knee injuries, but also obesity(increased body mass index(BMI)) ,joint malalignment and instability that result in increased mechanical stress are all strong risk factors for the development of knee OA [8-10].

Magnetic resonance imaging (MRI), arthroscopy examination, high-frequency color ultrasound and thermal texture maps are the four most acceptable types of imaging examinations. These examinations cannot only help diagnose KOA, but they can also assess the severity of joint damage and evaluate disease progression and treatment [11,12].

Treatment options for patients with OA include: conservative approaches, such as weight loss, physical therapy, and pharmacological interventions, while the more invasive approaches include intraarticular injections, joint preserving surgical treatment, and total knee arthroplasty (TKA). [13, 14] Radiofrequency ablation (RFA) is a novel technique that also recently gained popularity in alleviating chronic pain in patients with musculoskeletal disorders such as OA [15] Radiofrequency (RF) ablation, or modulation of the sensory innervation surrounding the knee, specifically the genicular nerves (GNs), has emerged as a therapeutic option to treat chronic knee OA pain for patients who are unresponsive to conservative treatments or are unsuitable candidates for total knee arthroplasty (TKA). [16, 17] In the case of knee OA, RFA was first introduced in 2010 by Choi et al and further explored in subsequent years [18,19] The mechanism of action of the therapy is that the RF lesion is believed to stop nociceptive (A-δ and C-fibers) pain input from the periphery to the central nervous system without destroying the motor or sensory (A-β) fibers. [15] More specifically, the postulated mechanism of action for clinical benefit of RFA involves the heat generation resulting in thermocoagulation and localized neuronal tissue destruction. These lesions have been shown to demonstrate the characteristics of scar formation, including an acute inflammatory response, cell necrosis, and fibrosis with collagen fiber deposition, occurring over 3 weeks following the procedure. It has been shown that the basal lamina of Schwann cells may be preserved after RFA, which would allow nerve regeneration. The threshold for neuronal tissue destruction has been shown to be 45°C in several studies . [15,24,25] Additionally, RFA produces a local electrical field, which is thought to promote neuromodulation by inhibition of the excitatory c-fibers. [25,26]

Similar to conventional RFA, water-cooled radiofrequency (CRF) ablation is a novel technology that utilizes thermal ablative mechanisms; however, CRF gives the ability to create a greater local neuronal lesion to increase the changes of effective denervation [20] In CRF, water circulates inside the probe to remove heat, modulating the thermal heat in the tissue to around 60°C, and alters the overall size, shape, and projections of lesions compared to conventional RFA. It is postulated that the greater sized CRF lesions may reduce the number of technical failures in the setting of a complex and variable neuronal innervation to the knee. The ability to target a greater amount of neuronal tissue is believed to produce long-term pain relief at least to the duration of relief produced by conventional RFA [27] A key limitation regarding standard RF techniques relates to the charring of tissues at the electrode interface. [28,29] Extended periods of ionic heating will cause desiccation and subsequent charring of the tissues immediately adjacent to the probe, as this tissue is absorbing the highest concentration of energy. Once the tissue becomes charred, it acts as a signiﬁcant insulator, preventing any subsequent energy moving beyond the charred tissue, limiting the size of lesions when standard RF technology is used Because of the size and shape limitations associated with standard RF ablation, it can be difﬁcult to reach the desired nerve target [30] In order to overcome the charring and subsequent insulation associated with standard RF, cooled radiofrequency probes were developed, whereby cooled water is circulated through the probe tip to maintain lower temperatures at the tissue-tip interface.

The circulated water serves to carry the heat away from the tissue-tip interface, which will reduce the desiccation and subsequent charring of adjacent tissues. As such, CRFA is able to deliver more energy to the surrounding tissues, creating a larger area where ionic heating can occur.

Relevant Anatomy Neuronal innervation of the knee is substantially intricate. The knee is innervated by the articular branches, known as the genicular nerves, of several major nerves, including the femoral, tibial, common peroneal (fibular), saphenous, and obturator nerves [21, 22] More specifically, the tibial nerve provides branches that innervate the articular capsule as they follow the superior medial and superior lateral vascular supplies [22,23] In the same way, the common peroneal nerve provides 2 articular branches that innervate the inferolateral articular capsule, while another common peroneal branch innervates the anterolateral as it follows the interior lateral genicular vasculature [22, 23] Thus, RFA requires identification of anatomical landmarks around the knee to locate the various genicular nerve branches that innervate the joint. As a result, the superomedial, superolateral, and inferomedial genicular nerve branches are commonly targeted by their proximal relation to bony landmarks . [18, 23]

ELIGIBILITY:
Inclusion Criteria:

* Patients with intractable knee pain intensity >5 on an 11-point visual analog scale (VAS) (where 0=no pain and 10=worst pain imaginable) for longer than three months and unable to do knee replacement surgery.
* Age > 50 years.
* Grade 2 or 3 KOA based on the Kellgren-Lawrence classification.
* Patients who did not respond to conservative treatment (physiotherapy, oral NSAIDs, and/or intraarticular injections of hyaluronic acid and corticosteroid) for 3 months.
* Duration of knee pain ≥ 3 months.
* Numeric rating scale (NRS) ≥ 5 points within 24 h prior to admission.

Exclusion Criteria:

* Grade 1 or 4 KOA based on the Kellgren-Lawrence classification.
* Severe liver, kidney, cardiovascular, and respiratory disease.
* Abnormal blood coagulation.
* Skin infections in the puncture region.
* Patients who previously underwent knee arthroscopy, TKA, RFTGN, or IAPRF.
* Mental disorders or inability to complete the follow-up observational form.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the ability to compare between cooled versus Thermocoagulant RF in the change from the baseline of the VAS for pain at the completion of treatment at 24 weeks. | 24weeks
  The primary outcome will be the ability to compare between cooled versus Thermocoagulant RF in the change from the baseline of the VAS for pain at the completion of treatment at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed MM Mostafa, A, professor, Study Director — Assiut University; Ahmed AA Abd elrahman, Doctor, Study Director — Assiut University